CLINICAL TRIAL: NCT06103396
Title: Treatment of Nonunion After Fractures (Pseudoartrosis) Using Mesenchymal Stromal Cells (MSCs)
Brief Title: Treatment of Nonunion Fractures With Mesenchymal Stromal Cells (MSCs)
Acronym: MSC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Venezolano de Investigaciones Cientificas (Other)
Collaborators: Hospital Central Dr. Plácido D. Rodriguez Rivero (Unknown); Instituto Autónomo Hospital Universitario de la Universidad de Los Andes (Unknown)
Responsible Party: Principal Investigator, Dylana Diaz Solano, Research Associate, Instituto Venezolano de Investigaciones Cientificas
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIC-UTC-MSC-Pseudarthrosis
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pseudoarthrosis of Bone; Pseudarthrosis; Non Union Fracture; Nonunion Bone Fracture
MeSH Terms: conditions — Pseudarthrosis; Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologuos MSCs transplantation in nonunion defects (Experimental): Autologuos MSCs harvested and cultured in osteogenic medium are seeded on collagen scaffold, and mixed with autologous rich plasma clot. The MSCs construct (MSCs/Col/PRP clot), is implanted in the nonunion defect.
  Interventions: Biological: Transplantation of autologous MSCs in nonunion fracture
- Allogeneic MSCs transplantation in nonunion defects (Experimental): Allogeneic MSCs harvested and cultured in osteogenic medium are seeded on collagen scaffold, and mixed with autologous rich plasma clot. The MSCs construct (MSCs/Col/PRP clot), is implanted in the nonunion defect.
  Interventions: Biological: Transplantation of allogeneic MSCs in nonunion fracture

INTERVENTIONS:
Biological: Transplantation of autologous MSCs in nonunion fracture — At surgery, fibrotic tissue is removed from the nonunion sites. MSCs/Col/PRP clots are implanted in the site of nonunion.
  Patients received conventional orthopedic treatment as they needed (osteotomy, external and/or internal fixation systems, etc.)
  Arms: Autologuos MSCs transplantation in nonunion defects
Biological: Transplantation of allogeneic MSCs in nonunion fracture — At surgery, fibrotic tissue is removed from the nonunion sites. MSCs/Col/PRP clots are implanted in the site of nonunion.
  Patients received conventional orthopedic treatment as they needed (osteotomy, external and/or internal fixation systems, etc.)
  Arms: Allogeneic MSCs transplantation in nonunion defects

SUMMARY:
The goal of this study is to evaluate the bone regeneration capacity of BM-MSC (Bone marrow mesenchymal stromal cells), in patients with nonunion. BM-MSC cultured are seeded on a collagen scaffold, included into autologous platelet-rich plasma (PRP) clot, and implanted in the nonunion bone defect.

DETAILED DESCRIPTION:
Nonunion (pseudoarthrosis) is one of the most serious complications of bone fracture. Even though different treatments have been used to repair nonunion bone defects, most of them have limitations, like morbidities, limited supply, frequent treatment failure, and high cost.

Based on the knowledge that MSC have multipotential capacity of differentiation into bone, cartilage, fat, and endothelial cells, and also, play a key role in the process of bone formation and fracture repair. In this study, we evaluated the use the bone regeneration capacity of autologous or allogeneic BM-MSC, as a potential therapeutic strategy to induce formation of new bone tissue and fracture healing.

A bioengineering construct, constituted by MSCs and a collagen scaffold, is incorporated into platelet rich plasma (PRP) clot, wich is implanted at the nonunion site defect.

ELIGIBILITY:
Inclusion Criteria:

* Post-traumatic nonunion diagnosis (Pseudoarthrosis) with or without previous ortopaedic treatment
* Patients with or without previous orthopaedic treatment
* Presence of nonunion 9 month or more
* Ossification failure in the non-union area, with an approximate size of 0.5 to 4 cm length

Exclusion Criteria:

* Evidence of infection at the nonunion site (Osteomielitis)
* Evidence of cutaneous lesion at the site of pseudoartrosis
* Viral hepatitis B and C, HIV infection, syphilis and other viral and bacterial infections
* Autoimmune diseases
* Neoplastic diseases
* Pregnancy
* Major metabolic disorders
* Treatment with steroids
* Other conditions or circumstances that compromise the study participation according to medical criteria

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | Baseline, 1 and 7 days. 1, 2 and 6 months. 1 and 2 years
  Time of surgical wound evolution, surgically intervened limb evolution, movility
Bone consolidation | Baseline, 1 and 7 days. 1, 2 and 6 months. 1 and 2 years
  Time of development changes in bone consolidation by radiological studies

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Cardier Montalvo, MD, PhD, Study Chair — Instituto Venezolano de Investigaciones Cientificas
Locations (1):
- Instituto Venezolano de Investigaciones Cientificas, Caracas, Miranda, Venezuela

REFERENCES:
- [Background] Wittig O, Romano E, Gonzalez C, Diaz-Solano D, Marquez ME, Tovar P, Aoun R, Cardier JE. A method of treatment for nonunion after fractures using mesenchymal stromal cells loaded on collagen microspheres and incorporated into platelet-rich plasma clots. Int Orthop. 2016 May;40(5):1033-8. doi: 10.1007/s00264-016-3130-6. Epub 2016 Mar 16. PMID 26980620
- [Background] Wittig O, Diaz-Solano D, Cardier J. Viability and functionality of mesenchymal stromal cells loaded on collagen microspheres and incorporated into plasma clots for orthopaedic application: Effect of storage conditions. Injury. 2018 Jun;49(6):1052-1057. doi: 10.1016/j.injury.2018.04.005. Epub 2018 Apr 5. PMID 29678307
- [Background] Diaz-Solano D, Wittig O, Mota JD, Cardier JE. Isolation and Characterization of Multipotential Mesenchymal Stromal Cells from Congenital Pseudoarthrosis of the Tibia: Case Report. Anat Rec (Hoboken). 2015 Oct;298(10):1804-14. doi: 10.1002/ar.23198. Epub 2015 Jul 30. PMID 26194170